CLINICAL TRIAL: NCT05681065
Title: Affective Based Integrated Care for Better Quality of Life (TeNDER).Pilot Implementation. Site 1: Primary Care Madrid, Spain.
Brief Title: Affective Based Integrated Care for Better Quality of Life.Pilot Implementation. Site1: Primary Care Madrid, Spain.
Acronym: TeNDER_Site1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Universidad Politecnica de Madrid (Other); Foundation for Biomedical Research and Innovation (Other)
Responsible Party: Principal Investigator, Cristina Lozano Hernández, Researcher on European projects. Family and Community Nurse Specialist, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 39/20; 875325 (Other Grant/Funding Number: Europe H2020)
Record Dates: First submitted 2023-01-03; First posted 2023-01-11 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Chronic Disease
Keywords: Chronic Disease; e-health; Quality of Life
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Design: randomised, open-label, multicentre, parallel-group clinical trial with 2-month follow-up.
  Patients in the intervention group will be fitted with the TeNDER system device best suited to the patient's needs, in addition to routine clinical practice. Patients in the control group will be treated according to standard clinical practice.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Standard practice. Patients will receive the usual clinical care based on the transmission of information and advice, and review according to the Clinical Practice Guidelines corresponding to the various chronic diseases presented by the patient.
- Intervention Group (Experimental): Standard practice. Patients will receive the usual clinical care based on the transmission of information and advice, and review according to the Clinical Practice Guidelines corresponding to the various chronic diseases presented by the patient. In addition, these participants will be provided with the TeNDER technological tool. The TeNDER intervention consists of the use of the TeNDER technological tool. It is a web application that integrates all the functionalities of the biosensors to facilitate patient self-monitoring, caregiver care and monitoring and management in the daily work of health professionals.
  Interventions: Device: TeNDER tool

INTERVENTIONS:
Device: TeNDER tool — The TeNDER intervention consists of the use of the TeNDER technological tool. It is a web application that integrates all the functionalities of biosensors to facilitate patient self-monitoring, caregiver care and monitoring and management in the daily work of healthcare professionals. Each participant will use the sensor that suits their needs:
  Sleep quality detector; Position sensor; Smart band; Smart watch; Microphone and speaker; rgb (real sense) sensor; Binary door and window sensor; Environmental sensor.
  Arms: Intervention Group

SUMMARY:
Objective: To evaluate the effectiveness of the TeNDER tool compared to usual practice in improving Quality of Life in patients with chronic diseases, according to type of disease and gender.

Methodology:

Design: randomised, open-label, multicentre, parallel-group clinical trial with 2-month follow-up.

Setting: health centres, homes, hospitals, socio-health centres and patient associations belonging to the participating countries.

Population: Patients with chronic diseases such as Parkinson's disease (PD), Alzheimer's disease or other dementias (AD) and cardiovascular disease (CVD); their caregivers and social-health professionals will be studied.

Sample size: n= 1,766 patients (1031 control/735 intervention).

Variables: The main outcome variable is the change in patient quality of life Short Form-36 Health Survey (SF-36). In addition, sociodemographic variables, technological affinity, usability, satisfaction and potential reductions in visits to health services after the intervention were collected in all study subjects. The change in patient autonomy after the intervention, the change in caregiver satisfaction with the care provided and the change in work overload in professionals were also studied.

Analysis: A descriptive analysis will be performed, a comparison of groups will be made at T1, a mean difference of global QoL and by dimensions will be calculated at T2 with its 95% Confident Interval (CI). For the main outcome, a multilevel linear regression model will be used with the dependent variable being the Quality of Life score at 60 days (T2) and the independent variable the group to which it belongs (control / TENDER) adjusted for possible confounding variables and/or effect modifiers. One model will be fitted for men and one for women. An intention-to-treat analysis will be performed.

DETAILED DESCRIPTION:
Hypothesis and Objective

Operational hypothesis: The use of the TeNDER tool by patients with chronic diseases increases their Quality of Life, as measured by the Short Form-36 Health Survey (SF-36), by at least 6 points, compared to usual practice.

Primary Aim: To evaluate the effectiveness of the TeNDER tool compared to usual practice in improving Quality of Life in patients with chronic diseases.

Secondary objectives:

* To evaluate the effectiveness of the TeNDER tool compared to usual practice in improving Quality of Life according to type of illness and gender.
* To evaluate the effectiveness of the TeNDER tool on caregiver overload.
* To describe the adherence and satisfaction of patients, carers and professionals with the TeNDER tool.

Methodology

Design: randomised, open-label, multicentre, parallel-group clinical trial with 2-month follow-up.

Patients in the intervention group will be fitted with the TeNDER system device best suited to the patient's needs, in addition to routine clinical practice. Patients in the control group will be treated according to standard clinical practice.

Sample size. The European consortium has proposed a sample size of 1766 patients (1031 in the Control Group and 735 in the Intervention Group). Those responsible for the technological development have considered that the tool will allow an improvement in Quality of Life (QoL) measured with the Short Form-36 Health Survey questionnaire of 6 points between the groups. According to previous studies consulted, the standard deviation of QoL in the population with the chronic diseases under study (PD, AD and CVD) varies between 16 and 27 [23-25]. For the power calculation, we have used the highest value of this standard deviation. Therefore, this sample size will allow a power of 98.8% to detect ≥6 differences in the overall score of the Short Form-36 Health Survey questionnaire if they exist.

The calculations were performed using a freely available software developed by public institutions for epidemiologists and other health professionals for the management of tabulated data.

In Primary Care of the Madrid Health Service, 534 patients will be included (380 in the Intervention Group and 254 in the Control Group). By pathology they will be: 80 patients with PD, 100 patients with AD and 360 patients with CVD.

Recruitment:

In each institution of the consortium, recruitment will be carried out according to its internal organisation.

For the Madrid Health Service institution, it is defined below:

Selection of centres and professionals: In Primary Care in Madrid, 5 health centres have been selected, including a total of 187 professionals (doctors and nurses) who will be offered to participate in the study. Based on experience in previous studies, we expect a participation rate of 45%, which means 84 participating professionals. If necessary, the number of participating centres will be expanded to reach the required sample size of patients and professionals.

Professionals will enter the study on a voluntary basis and after signing an informed consent form.

Recruitment of patients and carers:

Each participating professional will recruit 8 patients from their quota (5 with CVD, 1 with PD and 2 with AD). Recruitment will be done consecutively. Patients with some degree of dependence (PD and AD) will be recruited together with the caregiver, with the prior informed consent of both.

Participants must sign the informed consent before being included in the study. For this purpose, during the recruitment interview, the professionals will provide all the information about the study in written form and accompanied by a detailed verbal explanation, making sure that they understand it. You will be offered the information sheet to take home and share it with the people you consider important for the decision, at the same time as you will be offered the resolution of any doubts that may arise.

ELIGIBILITY:
The main study population is patients with Parkinson's disease (PD), Alzheimer's disease or other dementias (AD) and cardiovascular disease (CVD). Data will also be collected from their caregivers and professionals.

PATIENTS:

General Inclusion Criteria:

* Understand the local language of the country in which it takes place.
* Have a reference person or caregiver (if dependent).
* Agree to participate in the study, understand it and have signed the informed consent form.

Inclusion criteria for disease:

* AD: Persons expressing subjective cognitive compliant and Mini-Mental State Examination (MMSE) score of 19 to 28 pts, or having diagnosis of disease-causing dementia (with MMSE score of 19 to 28 pts) or Diagnosis of Alzheimer's according to National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
* PD: Confirmed diagnosis of Parkinson's disease. All patients will provide a report with an assessment from the neurologist.
* CVD: Patient that presents one of the following: cardiovascular failure grade II-III New York Heart Association (NYHA); coronary heart disease (both stable and acute coronary artery disease with or without S-T segment elevation); Atrial Fibrillation; Cardiac Pacemaker Carrier; Cerebral Stroke (ischaemic and haemorrhagic).

General Exclusion Criteria:

* Patients whose caregiver is not willing to participate / help; Patients / caregivers are not willing to work with the technologies used in this project.
* Patient and caregiver considered by the recruiting professional to be unable to follow the requirements of the study.
* Inability to move and move around at home (bedridden).
* Alcoholism or drug addiction.
* Life expectancy < 6 months.

Exclusion criteria for disease:

* AD: Advanced stages of the disease (GDS 6-7).
* PD: Parkinsonism secondary to vascular disease or treatment; Parkinsonism syndromes (Multiple System Atrophy, Progressive Supranuclear Palsy, Corticobasal Syndrome); dementia with Lewy bodies (DLB).
* CVD: acute coronary artery disease less than 4 weeks ago; severe aortic stenosis.

CAREGIVERS:

Inclusion criteria:

* To be able to consent and to comply with at least one of the following requisites:

  * To be employed by a public or private company or directly by the patients to provide direct care and thus support daily activities.
  * To live with and/or take care of a relative (or other close relationship) affected by Parkinson's disease or Alzheimer's disease or/and others forms of dementia or CVD
  * To provide logistic support to a family member or a close friend affected by Parkinson's disease or Alzheimer's disease or/and others forms of dementia or CVD.
* Express readiness in the use of technologies to use the devices

Exclusion criteria:

* Caregivers not able to consent.
* Caregivers not aware of the daily needs of patients.

PROFESSIONALS:

Inclusion criteria:

- To be able to consent and to be qualified and working in a medical or social area specialized in the care or support of persons with Parkinson's, Alzheimer's or/and other forms of dementia and cardiovascular diseases.

Exclusion criteria:

* Not working as a professional involved in the care or support of AD, PD, CVD patients.
* Working practice and environment not connected to Alzheimer's' and/or other forms of dementia, Parkinson's' disease or cardiovascular diseases.
* Conflict of interest.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in quality of life (PATIENT-ALL) | baseline and 1 month after intervention
  Quality of life will be measured at baseline and at the end of the TeNDER intervention (after 1 month) and the change between the two measures will be studied.
  Health-related quality of life as measured by the Short Form-36 Health Survey (SF-36). This questionnaire contains 36 items and 8 dimensions: Physical Function (10); Physical Role (4); Bodily Pain (2); General Health (5); Vitality (4); Social Function (2); Emotional Role (3) and 2 summary components (Physical and Mental).
  The score ranges from 0 to 100, where the higher the score the better the health status.

SECONDARY OUTCOMES:
Socio-demographic characteristics(PATIENT-ALL) | baseline
  Gender (male or female), age (number)
Main disease (PATIENT-ALL) | baseline
  Main disease shall be recorded as AD (Alzheimer disease, ) PD (Parkinson disease) and CVD (cardiovascular disease)
Technological affinity (PATIENT-ALL) | baseline
  This information is collected with a question about their taste for using technology and 6 different levels of response are offered.
Change in autonomy (PATIENT-ALL) | baseline and 1 month after intervention
  The difference in autonomy between baseline and after the intervention (1 month after) will be studied. Autonomy at each time point will be studied by means of 6 ad hoc likert-type questions scored 4-0. Where 24 is total autonomy and 0 is no autonomy.
Usability (PATIENT-INTERVENTION GROUP) | 1 month after intervention
  Collected through the validated tool "System Usability Scale". This scale is composed of 10 questions related to satisfaction with usability. The overall score is calculated from the sum of all item scores multiplied by 2.5, and the overall score ranges from 0 to 100.
Satisfaction (PATIENT-INTERVENTION GROUP) | 1 month after intervention
  Satisfaction with the intervention. This will be studied by means of 4 ad hoc likert-type questions scored 1-5. Where 20 is the highest satisfaction with the tool.
Potential reductions in visits to health services (PATIENT-INTERVENTION GROUP) | 1 month after intervention
  Through 3 questions, the opinion on the potential of the tool to reduce visits to health services is collected.

OTHER OUTCOMES:
Socio-demographic characteristics(CAREGIVERS) | baseline
  Gender (male or female), age (number)
Technological affinity(CAREGIVERS) | baseline
  This information is collected with a question about their taste for using technology and 6 different levels of response are offered.
Main disease on charge(CAREGIVERS) | baseline
  Main disease of the person being cared for. This shall be recorded as AD (Alzheimer disease, ) PD (Parkinson disease) and CVD (cardiovascular disease)
Change in quality of life (CAREGIVERS) | baseline and 1 month after intervention
  It will be collected through 11 ad hoc questions focused on the carer. It will be collected at baseline and 1 month after the intervention and the change will be studied.
Change in satisfaction with the care provided (CAREGIVERS) | baseline and 1 month after intervention
  By means of a question with different levels of response. It will be collected at baseline and 1 month after the intervention and the change will be studied.
Usability (CAREGIVERS) | 1 month after intervention
  Collected through the validated tool "System Usability Scale". This scale is composed of 10 questions related to satisfaction with usability. The overall score is calculated from the sum of all item scores multiplied by 2.5, and the overall score ranges from 0 to 100.
Satisfaction (CAREGIVERS) | 1 month after intervention
  Satisfaction with the intervention. This will be studied by means of 4 ad hoc likert-type questions scored 1-5. Where 20 is the highest satisfaction with the tool.
Potential reductions in visits to health services (CAREGIVERS) | 1 month after intervention
  Through 3 questions, the opinion on the potential of the tool to reduce visits to health services is collected.
Socio-demographic characteristics (PROFESSIONALS) | baseline
  Gender (male or female), age (number)
Technological affinity (PROFESSIONALS) | baseline
  This information is collected with a question about their taste for using technology and 6 different levels of response are offered.
Change in work overload (PROFESSIONALS) | baseline and 1 month after intervention
  By means of a question with different levels of response. It will be collected at baseline and 1 month after the intervention and the change will be studied.
Usability (PROFESSIONALS) | 1 month after intervention
  Collected through the validated tool "System Usability Scale". This scale is composed of 10 questions related to satisfaction with usability. The overall score is calculated from the sum of all item scores multiplied by 2.5, and the overall score ranges from 0 to 100.
Satisfaction (PROFESSIONALS) | 1 month after intervention
  Satisfaction with the intervention. This will be studied by means of 4 ad hoc likert-type questions scored 1-5. Where 20 is the highest satisfaction with the tool.
Potential reductions in visits to health services (PROFESSIONALS) | 1 month after intervention
  Through 3 questions, the opinion on the potential of the tool to reduce visits to health services is collected.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Álvarez, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Gerencia de atención primaria, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Violan C, Foguet-Boreu Q, Flores-Mateo G, Salisbury C, Blom J, Freitag M, Glynn L, Muth C, Valderas JM. Prevalence, determinants and patterns of multimorbidity in primary care: a systematic review of observational studies. PLoS One. 2014 Jul 21;9(7):e102149. doi: 10.1371/journal.pone.0102149. eCollection 2014. PMID 25048354
- [Background] Haslbeck J, Zanoni S, Hartung U, Klein M, Gabriel E, Eicher M, Schulz PJ. Introducing the chronic disease self-management program in Switzerland and other German-speaking countries: findings of a cross-border adaptation using a multiple-methods approach. BMC Health Serv Res. 2015 Dec 28;15:576. doi: 10.1186/s12913-015-1251-z. PMID 26711458
- [Background] Davis AA, Racette B. Parkinson disease and cognitive impairment: Five new things. Neurol Clin Pract. 2016 Oct;6(5):452-458. doi: 10.1212/CPJ.0000000000000285. PMID 27847686
- [Background] Mills SL, Brady TJ, Jayanthan J, Ziabakhsh S, Sargious PM. Toward consensus on self-management support: the international chronic condition self-management support framework. Health Promot Int. 2017 Dec 1;32(6):942-952. doi: 10.1093/heapro/daw030. PMID 27242377
- [Background] Ornstein SM, Nietert PJ, Jenkins RG, Litvin CB. The prevalence of chronic diseases and multimorbidity in primary care practice: a PPRNet report. J Am Board Fam Med. 2013 Sep-Oct;26(5):518-24. doi: 10.3122/jabfm.2013.05.130012. PMID 24004703
- [Background] Konig HH, Leicht H, Bickel H, Fuchs A, Gensichen J, Maier W, Mergenthal K, Riedel-Heller S, Schafer I, Schon G, Weyerer S, Wiese B, Bussche Hv, Scherer M, Eckardt M; MultiCare study group. Effects of multiple chronic conditions on health care costs: an analysis based on an advanced tree-based regression model. BMC Health Serv Res. 2013 Jun 15;13:219. doi: 10.1186/1472-6963-13-219. PMID 23768192
- [Background] Torous J, Kiang MV, Lorme J, Onnela JP. New Tools for New Research in Psychiatry: A Scalable and Customizable Platform to Empower Data Driven Smartphone Research. JMIR Ment Health. 2016 May 5;3(2):e16. doi: 10.2196/mental.5165. PMID 27150677
- [Background] Mohr DC, Zhang M, Schueller SM. Personal Sensing: Understanding Mental Health Using Ubiquitous Sensors and Machine Learning. Annu Rev Clin Psychol. 2017 May 8;13:23-47. doi: 10.1146/annurev-clinpsy-032816-044949. Epub 2017 Mar 17. PMID 28375728
- [Background] Raggi A, Corso B, Minicuci N, Quintas R, Sattin D, De Torres L, Chatterji S, Frisoni GB, Haro JM, Koskinen S, Martinuzzi A, Miret M, Tobiasz-Adamczyk B, Leonardi M. Determinants of Quality of Life in Ageing Populations: Results from a Cross-Sectional Study in Finland, Poland and Spain. PLoS One. 2016 Jul 19;11(7):e0159293. doi: 10.1371/journal.pone.0159293. eCollection 2016. PMID 27434374
- [Background] Huckvale K, Venkatesh S, Christensen H. Toward clinical digital phenotyping: a timely opportunity to consider purpose, quality, and safety. NPJ Digit Med. 2019 Sep 6;2:88. doi: 10.1038/s41746-019-0166-1. eCollection 2019. PMID 31508498
- [Background] Kitsiou S, Pare G, Jaana M, Gerber B. Effectiveness of mHealth interventions for patients with diabetes: An overview of systematic reviews. PLoS One. 2017 Mar 1;12(3):e0173160. doi: 10.1371/journal.pone.0173160. eCollection 2017. PMID 28249025
- [Background] Tu XJ, Hwang WJ, Ma HI, Chang LH, Hsu SP. Determinants of generic and specific health-related quality of life in patients with Parkinson's disease. PLoS One. 2017 Jun 26;12(6):e0178896. doi: 10.1371/journal.pone.0178896. eCollection 2017. PMID 28650957
- [Background] Benda NM, Seeger JP, Stevens GG, Hijmans-Kersten BT, van Dijk AP, Bellersen L, Lamfers EJ, Hopman MT, Thijssen DH. Effects of High-Intensity Interval Training versus Continuous Training on Physical Fitness, Cardiovascular Function and Quality of Life in Heart Failure Patients. PLoS One. 2015 Oct 30;10(10):e0141256. doi: 10.1371/journal.pone.0141256. eCollection 2015. PMID 26517867
- [Background] Geschke K, Fellgiebel A, Laux N, Schermuly I, Scheurich A. Quality of life in dementia: impact of cognition and insight on applicability of the SF-36. Am J Geriatr Psychiatry. 2013 Jul;21(7):646-54. doi: 10.1016/j.jagp.2012.12.014. Epub 2013 Feb 6. PMID 23567410
- [Background] Vilagut G, Ferrer M, Rajmil L, Rebollo P, Permanyer-Miralda G, Quintana JM, Santed R, Valderas JM, Ribera A, Domingo-Salvany A, Alonso J. [The Spanish version of the Short Form 36 Health Survey: a decade of experience and new developments]. Gac Sanit. 2005 Mar-Apr;19(2):135-50. doi: 10.1157/13074369. Spanish. PMID 15860162
- [Background] Perera R, Heneghan C, Yudkin P. Graphical method for depicting randomised trials of complex interventions. BMJ. 2007 Jan 20;334(7585):127-9. doi: 10.1136/bmj.39045.396817.68. PMID 17235093
- [Derived] Medina-Garcia R, Lopez-Rodriguez JA, Lozano-Hernandez CM, Ruiz Bejerano V, Criscio P, Del Cura-Gonzalez I; TeNDER Atencion Primaria Group. A Technological Tool Aimed at Self-Care in Patients With Multimorbidity: Cross-Sectional Usability Study. JMIR Hum Factors. 2024 Apr 5;11:e46811. doi: 10.2196/46811. PMID 38578675
- [Derived] Lozano Hernandez CM, Medina-Garcia R, de Hoyos-Alonso MC, Garrido-Barral A, Minue Lorenzo C, Sanz-Cuesta T, Serrano J, Del Rio Ponce A, Gomez-Gascon T, Del Cura-Gonzalez I; TeNDER Group Primary Care. Improvement in Quality of Life With the Use of a Technological System Among Patients With Chronic Disease Followed Up in Primary Care (TeNDER Project): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Jul 3;12:e47331. doi: 10.2196/47331. PMID 37399054
- See also: World Health Organization (WHO) apps website — http://apps.who.int/iris/
- See also: World Health Organization (WHO) website — https://www.who.int/es/news-room/fact-sheets/detail/cardiovascular-diseases-(cvds)